CLINICAL TRIAL: NCT04396691
Title: Clinimetric and Instrumental Characterization of Fighter Pilots With Flight-related Neck Pain. Observational Study
Brief Title: Clinimetric and Instrumental Characterization of Fighter Pilots With Flight-related Neck Pain.
Status: Completed | Type: Observational
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Carlos Fernández-Morales, PT, MSc, Universidad de Extremadura
Other Study IDs: 01
Record Dates: First submitted 2020-05-19; First posted 2020-05-20 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Neck Pain
Keywords: nonspecific chronic neck pain; fighter pilots
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Instructors group: Group of flight instructors at the reactor school.
- Students group: Group of students at the reactor school.

SUMMARY:
The objective of the study is to detect the state of clinical and instrumental factors related in fighter pilots with non-specific mechanical neck pain.

DETAILED DESCRIPTION:
A prevalence study (descriptive, observational, cross-sectional) was carried out, in which clinimetric variables (range of active cervical movement, motor control and electrical activity), perceived pain (using NSMNP and algometry) and disability were evaluated. The sample (n = 18) is divided into instructors (n = 7) and students (n = 11). The objective of this study is to characterize descriptively at the sociodemographic level and to know the state of health in relation to clinimetric variables of the fighter pilots of the Talavera la Real air base (Badajoz) to determine the risk of developing an neck injury.

ELIGIBILITY:
Inclusion Criteria:

* Numerical pain rating scale. Participants rated the intensity of their neck pain at rest on an 11-point Numeric Pain Rating Scale (NPRS), where 0 was no pain and 10 maximum pain .The pilots airforce were asked to indicate the pain levels that they experienced when they wake up in the morning. Cleland et al reported that the minimal detectable change (MDC) and minimal clinically important difference (MCID) for the numeric pain rating scale were 1.3 and 2.1 points, respectively, in patients with mechanical neck pain.
* Joint Position Sense. This test assesses the ability to relocate the head to its natural posture, and is a test of cervical proprioception. It consists of a visual measurement of error in moving the head to the initial neutral position after active cervical rotation. If the average difference between the initial and final position is equivalent to an error of 4.5 degrees, it is considered abnormal and the subject could be included in the study.

Exclusion Criteria:

* Cervical pain that occurs with irradiation to the upper limbs and / or radiculopathy.
* Cervical spine surgery.
* Have received physical therapy treatment six weeks prior to data collection.
* Being involved in an on-going medico-legal dispute.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The selection of the sample was made in the accessible population of the Talavera la Real Air Base (Badajoz).
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Range of movement | 1 week
  For the evaluation of cervical ROM, we will use a conventional two-branch goniometer, from the EnrafNonius® brand. Subjects will be placed in a sitting position on a stool, with a neutral neck and head position. The range of active cervical mobility presented by the patients was measured in reference to the three planes of the space. In the sagittal plane, the degrees of mobility to flexion and extension were measured, in the frontal plane the right and left inclinations, and in the transverse plane both rotations.
Disability | 1 week
  The degree of cervical disability involvement was measured through the Neck Disability Index (NDI), translated into Spanish, presenting optimum reliability and internal validity. It consists of 10 sections, 4 of them are related to subjective symptoms and the other 6 are related to basic activities of daily life.
  Each of the sections presents 6 possible responses, scoring these from 0 to 5 according to progression of functional disability.
  Scores less than 5 points indicate non-disability, between 5-14 points indicates mild disability, values between 30-48 points moderate disability, between 50-64 points severe disability and those that exceed 70 points represent complete disability.

SECONDARY OUTCOMES:
Pressure pain thresholds | 1 week
  A mechanical pressure Fisher algometer (Force Dial model FDK 40) with a 1 cm² area contact head was used to measure the pressure pain threshold. The reliability of pressure algometry has been found to be high [intraclass correlation coefficient = 0.91 (95% confidence interval, 0.82-0.97)]. With the participant in supine, the pressure pain threshold of the the myofascial trigger point nº2 of the upper trapezius muscle according to Travell and Simons and the central trigger point of the sternocleidomastoid muscle was bilaterally evaluated. Also, in sitting position the pressure pain threshold of the myofascial trigger point of the scapula elevator muscle was bilaterally evaluated. The minimal clinically important difference (MCDI) is 1.2 Kg/cm2.
Surface electromyographic | 1 week
  The electromyography (EMG) signal of the upper trapezius muscle was recorded during 3 step contractions of shoulder elevation force (15%-30% maximal voluntary contraction). Se tomo el valor más alto de las tres contracciones. The signal of the sternocleidomastoid muscle was recorded during 3 billateraly step contractions of neck flexión and antepulsion neck force. Both contractions were performed in a combined and simultaneous movement, recreating the movement produced by the reaction forces in the takeoff and landing of the fighter jet. Both movements were made at 15%-30% maximal voluntary contraction, as used by Calamita et al on the same musculature in subjects with nonspecific neck pain.
Kinesophobia | 1 week
  The Spanish version of the TSK-11 was used to measure fear of movement. Higher scores indicate greater fear-avoidance behaviors. The TSK-11 has demonstrated acceptable internal consistency and validity.
Catastrophic pain | 1 week
  The Pain Catastrophizing Scale (PCS) is a self-administered scale of 13 items and one of the most used to assess catastrophism of pain. The subjects take their past painful experiences as a reference and indicate the degree to which they experienced each of the 13 thoughts or feelings on a 5-point Líkert scale ranging from 0 (never) to 4 (always). The theoretical range of the instrument is between 13 and 62, indicating low scores, little catastrophism, and high values, high catastrophism.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Fernández-Morales, PT, MSc, Principal Investigator — Universidad de Extremadura
Locations (1):
- Universidad de Extremadura, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jensen MP, Turner JA, Romano JM, Fisher LD. Comparative reliability and validity of chronic pain intensity measures. Pain. 1999 Nov;83(2):157-62. doi: 10.1016/s0304-3959(99)00101-3. PMID 10534586
- [Background] Cleland JA, Childs JD, Whitman JM. Psychometric properties of the Neck Disability Index and Numeric Pain Rating Scale in patients with mechanical neck pain. Arch Phys Med Rehabil. 2008 Jan;89(1):69-74. doi: 10.1016/j.apmr.2007.08.126. PMID 18164333
- [Background] Chesterton LS, Sim J, Wright CC, Foster NE. Interrater reliability of algometry in measuring pressure pain thresholds in healthy humans, using multiple raters. Clin J Pain. 2007 Nov-Dec;23(9):760-6. doi: 10.1097/AJP.0b013e318154b6ae. PMID 18075402
- [Background] Hapidou EG, O'Brien MA, Pierrynowski MR, de Las Heras E, Patel M, Patla T. Fear and Avoidance of Movement in People with Chronic Pain: Psychometric Properties of the 11-Item Tampa Scale for Kinesiophobia (TSK-11). Physiother Can. 2012 Summer;64(3):235-41. doi: 10.3138/ptc.2011-10. PMID 23729957
- [Background] Gomez-Perez L, Lopez-Martinez AE, Ruiz-Parraga GT. Psychometric Properties of the Spanish Version of the Tampa Scale for Kinesiophobia (TSK). J Pain. 2011 Apr;12(4):425-35. doi: 10.1016/j.jpain.2010.08.004. PMID 20926355
- [Background] Calamita SAP, Biasotto-Gonzalez DA, De Melo NC, Fumagalli MA, Amorim CF, de Paula Gomes CAF, Politti F. Immediate Effect of Acupuncture on Electromyographic Activity of the Upper Trapezius Muscle and Pain in Patients With Nonspecific Neck Pain: A Randomized, Single-Blinded, Sham-Controlled, Crossover Study. J Manipulative Physiol Ther. 2018 Mar-Apr;41(3):208-217. doi: 10.1016/j.jmpt.2017.09.006. PMID 29549891
- [Background] Sullivan MJ, Bishop SR, Pivik J. The pain catastrophizing scale: development and validation. Psychol Assess. 1995;7(4):524.
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Background] Peterson-Kendall F, Kendall-McCreary E, Geise-Provance P, McIntyre-Rodgers M, Romani W. Muscles testing and function with posture and pain. US Lippincott Williams Wilkins Ltd. 2005;49-118.
- [Background] MacDermid JC, Walton DM, Avery S, Blanchard A, Etruw E, McAlpine C, Goldsmith CH. Measurement properties of the neck disability index: a systematic review. J Orthop Sports Phys Ther. 2009 May;39(5):400-17. doi: 10.2519/jospt.2009.2930. PMID 19521015
- [Background] Kovacs FM, Bago J, Royuela A, Seco J, Gimenez S, Muriel A, Abraira V, Martin JL, Pena JL, Gestoso M, Mufraggi N, Nunez M, Corcoll J, Gomez-Ochoa I, Ramirez MJ, Calvo E, Castillo MD, Marti D, Fuster S, Fernandez C, Gimeno N, Carballo A, Milan A, Vazquez D, Canellas M, Blanco R, Brieva P, Rueda MT, Alvarez L, Del Real MT, Ayerbe J, Gonzalez L, Ginel L, Ortega M, Bernal M, Bolado G, Vidal A, Ausin A, Ramon D, Mir MA, Tomas M, Zamora J, Cano A. Psychometric characteristics of the Spanish version of instruments to measure neck pain disability. BMC Musculoskelet Disord. 2008 Apr 9;9:42. doi: 10.1186/1471-2474-9-42. PMID 18400084
- [Background] Revel M, Andre-Deshays C, Minguet M. Cervicocephalic kinesthetic sensibility in patients with cervical pain. Arch Phys Med Rehabil. 1991 Apr;72(5):288-91. PMID 2009044